CLINICAL TRIAL: NCT06662929
Title: Arabic Patient-reported Outcome Measures During Radiotherapy for Head and Neck Cancer: a Validation Study
Brief Title: Arabic PRO Measures for Head and Neck Cancer Radiotherapy.
Acronym: PROMs
Status: Recruiting | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Abdullah Mohamed Alsoghier, PhD, Consultant, Assistant Professor, King Saud University
Other Study IDs: E-23-7571
Record Dates: First submitted 2023-10-19; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms; Head and Neck Squamous Cell Carcinoma; Oropharynx Cancer; Nasopharyngeal Cancer; Oral Cancer; Tongue Cancer; Oral Neoplasm
Keywords: PROMs; Head and Neck Cancer; Radiotherapy; COSMIN; Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Nasopharyngeal Neoplasms; Mouth Neoplasms; Tongue Neoplasms; Neoplasms | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult aged 18 years or above, and receiving radiotherapy for the HNC.: A non-interventional, questionnaire-based cross-sectional study for Arabic-speaking males and females, aged 18 years or above who is planned for receiving and who is currently receiving and who had already received radiotherapy for the Head & Neck Cancer at King Saud University Medical City.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiotherapy for the Head & Neck Cancer

SUMMARY:
The goal of Arabic patient-reported outcome measures during radiotherapy for head and neck cancer is to test the patient-reported outcome measure (PROM) tools. PROM tools are not validated cross-culturally in Arabic-speaking patient populations, which limits their use in our clinical setting. Validation of these PROM tools will allow clinicians to identify the concerns related to our patient population and measure the outcome of our interventions. Main objectives are:

* To further validate (cross-culture) the PROM instruments related to head and neck cancer (HNC) in Arabic patients.
* To investigate the prevalence and severity of the patient-reported concerns and their relevance with demographics and clinical characteristics.

The participants will be given tasks to complete 6 tools survey before, during, and after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or above and who is planned for receiving and who is currently receiving and who had already received radiotherapy for the HNC at King Saud University Medical City.

Exclusion Criteria:

* Individuals who are less than 18 years, presence of debilitating disease (e.g. heart failure) or who lack the capacity to read, understand and sign the informed consent and those.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target Population: The study is targeting males and females aged 18 years or above, and receiving radiotherapy for the HNC at the King Saud University Medical City.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Summated Xerostomia Inventory (SXI) | 24 months
  The study aimed to assess the validity (face, content and construct) and reliability (internal consistency and test-retest) of this inventory in patients who received radiotherapy for head and neck cancer. These will be conducted in line with COnsensus-based Standards for the selection of health Measurement INstruments (COSMIN) guidelines.
Patient-Reported Oral Mucositis Symptom (PROM) scale | 24 months
  The study aimed to assess the validity (face, content and construct) and reliability (internal consistency and test-retest) of this inventory in patients who received radiotherapy for head and neck cancer. These will be conducted in line with COnsensus-based Standards for the selection of health Measurement INstruments (COSMIN) guidelines.
The Arabic University of Washington questionnaire (UW-QOL v4) | 24 months
  The study aimed to assess the validity (face, content and construct) and reliability (internal consistency and test-retest) of this inventory in patients who received radiotherapy for head and neck cancer. These will be conducted in line with COnsensus-based Standards for the selection of health Measurement INstruments (COSMIN) guidelines.
The Arabic Brief Fatigue Inventory (ArBFI) | 24 months
  The study aimed to assess the validity (face, content and construct) and reliability (internal consistency and test-retest) of this inventory in patients who received radiotherapy for head and neck cancer. These will be conducted in line with COnsensus-based Standards for the selection of health Measurement INstruments (COSMIN) guidelines.
Patient Concerns Inventory - Head and Neck (PCI-HNC) | 24 months
  The study aimed to assess the validity (face, content and construct) and reliability (internal consistency and test-retest) of this inventory in patients who received radiotherapy for head and neck cancer. These will be conducted in line with COnsensus-based Standards for the selection of health Measurement INstruments (COSMIN) guidelines.

SECONDARY OUTCOMES:
To investigate the prevalence and severity of the patient-reported concerns and their relevance with demographics and clinical characteristics. | 24 months
  Descriptive statistics [frequencies with percentage (%) for categorical variables, and the mean (±SD) and median for numerical variables collected] will be used to for patients' demographic and clinical characteristics and study measures using SPSS v.22 (IBM, Armonk, New York). Level of significance will be set at or below 0.05. Correlations between study findings will be assessed using Pearson or Spearman's correlation coefficients - based on normality of data. Regression analyses for patient characteristics and measurement variables.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aguilar ML, Sandow P, Werning JW, Brenneman L, Psoter WJ. The Head and Neck Cancer Patient Concern Inventory(c) : Patient Concerns' Prevalence, Dental Concerns' Impact, and Relationships of Concerns with Quality of Life Measures. J Prosthodont. 2017 Apr;26(3):186-195. doi: 10.1111/jopr.12496. Epub 2017 Feb 21. PMID 28220985
- [Background] Alhazzazi TY, Alghamdi FT. Head and Neck Cancer in Saudi Arabia: a Systematic Review. Asian Pac J Cancer Prev. 2016;17(8):4043-8. PMID 27644659
- [Background] Alqaryan S, Aldrees T, Almatrafi S, Alharbi A, Alhumaid H. Awareness of head and neck cancers in Saudi Arabia. A questionnaire based study. Saudi Med J. 2020 Apr;41(4):400-405. doi: 10.15537/smj.2020.4.24990. PMID 32291427
- [Background] Berger AM, Abernethy AP, Atkinson A, Barsevick AM, Breitbart WS, Cella D, Cimprich B, Cleeland C, Eisenberger MA, Escalante CP, Jacobsen PB, Kaldor P, Ligibel JA, Murphy BA, O'Connor T, Pirl WF, Rodler E, Rugo HS, Thomas J, Wagner LI. NCCN Clinical Practice Guidelines Cancer-related fatigue. J Natl Compr Canc Netw. 2010 Aug;8(8):904-31. doi: 10.6004/jnccn.2010.0067. No abstract available. PMID 20870636
- [Background] Black N. Patient reported outcome measures could help transform healthcare. BMJ. 2013 Jan 28;346:f167. doi: 10.1136/bmj.f167. PMID 23358487
- [Background] Catania G, Bell C, Ottonelli S, Marchetti M, Bryce J, Grossi A, Costantini M. Cancer-related fatigue in Italian cancer patients: validation of the Italian version of the Brief Fatigue Inventory (BFI). Support Care Cancer. 2013 Feb;21(2):413-9. doi: 10.1007/s00520-012-1539-z. Epub 2012 Jul 13. PMID 22790224
- [Background] Cruz FM, Munhoz BA, Alves BC, Gehrke FS, Fonseca FL, Kuniyoshi RK, Cubero D, Peppone LJ, Del Giglio A. Biomarkers of fatigue related to adjuvant chemotherapy for breast cancer: evaluation of plasma and lymphocyte expression. Clin Transl Med. 2015 Feb 14;4:4. doi: 10.1186/s40169-015-0051-8. eCollection 2015. PMID 25852820
- [Background] Dirix P, Nuyts S, Van den Bogaert W. Radiation-induced xerostomia in patients with head and neck cancer: a literature review. Cancer. 2006 Dec 1;107(11):2525-34. doi: 10.1002/cncr.22302. PMID 17078052
- [Background] Hamilton SN, Tran E, Ho C, Berthelet E, Wu J, DeVries K, LaPointe V, Bowman A, Lagman M, Olson R. Patient-reported outcome measures in patients undergoing radiotherapy for head and neck cancer. Support Care Cancer. 2021 May;29(5):2537-2547. doi: 10.1007/s00520-020-05778-2. Epub 2020 Sep 19. PMID 32949298
- [Background] Kanatas A, Lowe D, Rogers SN. Health-related quality of life at 3 months following head and neck cancer treatment is a key predictor of longer-term outcome and of benefit from using the patient concerns inventory. Cancer Med. 2022 Apr;11(8):1879-1890. doi: 10.1002/cam4.4558. Epub 2022 Feb 17. PMID 35178880
- [Background] Kingsley C, Patel S. Patient-reported outcome measures and patient-reported experience measures. BJA Education. 2017;17(4):137-44.
- [Background] Kushner JA, Lawrence HP, Shoval I, Kiss TL, Devins GM, Lee L, Tenenbaum HC. Development and validation of a Patient-Reported Oral Mucositis Symptom (PROMS) scale. J Can Dent Assoc. 2008 Feb;74(1):59. PMID 18298885
- [Background] Mehanna H, Paleri V, West CM, Nutting C. Head and neck cancer--Part 1: Epidemiology, presentation, and prevention. BMJ. 2010 Sep 20;341:c4684. doi: 10.1136/bmj.c4684. No abstract available. PMID 20855405
- [Background] Mody MD, Rocco JW, Yom SS, Haddad RI, Saba NF. Head and neck cancer. Lancet. 2021 Dec 18;398(10318):2289-2299. doi: 10.1016/S0140-6736(21)01550-6. Epub 2021 Sep 22. PMID 34562395
- [Background] Okuyama T, Wang XS, Akechi T, Mendoza TR, Hosaka T, Cleeland CS, Uchitomi Y. Validation study of the Japanese version of the brief fatigue inventory. J Pain Symptom Manage. 2003 Feb;25(2):106-17. doi: 10.1016/s0885-3924(02)00596-1. PMID 12590026
- [Background] Rogers SN, El-Sheikha J, Lowe D. The development of a Patients Concerns Inventory (PCI) to help reveal patients concerns in the head and neck clinic. Oral Oncol. 2009 Jul;45(7):555-61. doi: 10.1016/j.oraloncology.2008.09.004. Epub 2008 Nov 22. PMID 19028135
- [Background] Senkal HA, Hayran M, Karakaya E, Yueh B, Weymuller EA Jr, Hosal AS. The validity and reliability of the Turkish version of the University of Washington Quality of Life Questionnaire for patients with head and neck cancer. Am J Otolaryngol. 2012 Jul-Aug;33(4):417-26. doi: 10.1016/j.amjoto.2011.10.014. Epub 2011 Dec 1. PMID 22137146
- [Background] Sharour LA. Translation and Validation of the Arabic Version of the Cancer Needs Questionnaire-Short Form. Asia Pac J Oncol Nurs. 2020 Oct 15;8(1):74-80. doi: 10.4103/apjon.apjon_33_20. eCollection 2021 Jan-Feb. PMID 33426193
- [Background] Sroussi HY, Epstein JB, Bensadoun RJ, Saunders DP, Lalla RV, Migliorati CA, Heaivilin N, Zumsteg ZS. Common oral complications of head and neck cancer radiation therapy: mucositis, infections, saliva change, fibrosis, sensory dysfunctions, dental caries, periodontal disease, and osteoradionecrosis. Cancer Med. 2017 Dec;6(12):2918-2931. doi: 10.1002/cam4.1221. Epub 2017 Oct 25. PMID 29071801
- [Background] Thomson WM, van der Putten GJ, de Baat C, Ikebe K, Matsuda K, Enoki K, Hopcraft MS, Ling GY. Shortening the xerostomia inventory. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Sep;112(3):322-7. doi: 10.1016/j.tripleo.2011.03.024. Epub 2011 Jul 16. PMID 21684773
- [Background] Vartanian JG, Carvalho AL, Yueh B, Priante AV, de Melo RL, Correia LM, Kohler HF, Toyota J, Kowalski IS, Kowalski LP. Long-term quality-of-life evaluation after head and neck cancer treatment in a developing country. Arch Otolaryngol Head Neck Surg. 2004 Oct;130(10):1209-13. doi: 10.1001/archotol.130.10.1209. PMID 15492171
- [Background] Wijers OB, Levendag PC, Braaksma MM, Boonzaaijer M, Visch LL, Schmitz PI. Patients with head and neck cancer cured by radiation therapy: a survey of the dry mouth syndrome in long-term survivors. Head Neck. 2002 Aug;24(8):737-47. doi: 10.1002/hed.10129. PMID 12203798
- [Background] Mokkink LB, Terwee CB, Knol DL, Stratford PW, Alonso J, Patrick DL, Bouter LM, de Vet HC. The COSMIN checklist for evaluating the methodological quality of studies on measurement properties: a clarification of its content. BMC Med Res Methodol. 2010 Mar 18;10:22. doi: 10.1186/1471-2288-10-22. PMID 20298572
- [Background] Gagnier JJ, Lai J, Mokkink LB, Terwee CB. COSMIN reporting guideline for studies on measurement properties of patient-reported outcome measures. Qual Life Res. 2021 Aug;30(8):2197-2218. doi: 10.1007/s11136-021-02822-4. Epub 2021 Apr 5. PMID 33818733
- [Background] Suleiman K, Al Kalaldeh M, AbuSharour L, Yates B, Berger A, Mendoza T, Malak M, Salameh AB, Cleeland C, Menshawi A. Validation study of the Arabic version of the Brief Fatigue Inventory (BFI-A). East Mediterr Health J. 2019 Nov 25;25(11):784-790. doi: 10.26719/emhj.19.032. PMID 31782514